CLINICAL TRIAL: NCT05625009
Title: Comparison of Bilateral Ultrasound-Guided Transversus Abdominis Plane (Tap) Block and Erector Spinal Plane (Esp) Block in the Management of Postoperative Analgesia in Patients Who Had Cesarean Section Under Spinal Anesthesia
Brief Title: Bilateral Ultrasound-Guided Transversus Abdominis Plane (Tap) Block and Erector Spinal Plane (Esp) Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Taner Abdullah, Principal Investigator, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021.10.227
Record Dates: First submitted 2022-11-11; First posted 2022-11-22 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Pain, Postoperative; Cesarean Section; Erector Spinae Plane Block; Transversus Abdominis Plane Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators who assessed pain scores postoperatively are blinded to the study groups Care providers on the yard are blinded to the study groups Outcome assessors are blinded to the study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Transversus Abdominis Plane Block (TAPB) (Experimental): patients received TAPB postoperatively
  Interventions: Procedure: Procedure/Surgery: Transversus Abdominis Plane Block (TAPB)
- Experimental: Erector Spinae Plane Block (ESPB) (Experimental): patients received ESPB postoperatively
  Interventions: Procedure: Procedure/Surgery: Erector Spinae Plane Block (ESPB)

INTERVENTIONS:
Procedure: Procedure/Surgery: Transversus Abdominis Plane Block (TAPB) — Patients received TAPB postoperatively
  Arms: Experimental: Transversus Abdominis Plane Block (TAPB)
Procedure: Procedure/Surgery: Erector Spinae Plane Block (ESPB) — Patients received ESPB postoperatively
  Arms: Experimental: Erector Spinae Plane Block (ESPB)

SUMMARY:
Transversus Abdominis Plane Block (TAPB) is frequently used for the management of postoperative pain in patients undergoing cesarean section. Recently, Erector Spinae Plane Block (ESPB) has been defined and used in several clinical scenarios. However, data regarding the ESPB use in the aforementioned patient group is limited.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 45 years
* ASA2
* Undergoing cesarean section under spinal anesthesia

Exclusion Criteria:

* History of chronic pain
* Body mass index > 35
* Urgent/emergent surgeries
* Major bleeding
* Any additional surgical procedure
* Contraindication for any drugs used in the protocol
* The presence of any instrumentation in the procedure sites

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — cesarean section
Enrollment: 94 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients needed for rescue analgesic agent (diclofenac) | 24 hours

SECONDARY OUTCOMES:
Percentage of patients needed for rescue analgesic agent (opioid) | 24 hours
the dose of the opioid used | 24 hours
Percentage of patients experienced chronic pain | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Basaksehir Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes